CLINICAL TRIAL: NCT06410248
Title: A Phase 1 Adaptive Dose Escalation With Dose Expansion Study of Triapine in Combination With Temozolomide (TMZ) for Patients With Recurrent Glioblastoma
Brief Title: Triapine in Combination With Temozolomide for the Treatment of Patients With Recurrent Glioblastoma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH); BrainUp Inc (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NU 23C05; NCI-2024-02351 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STU00220426; NU 23C05 (Other: Northwestern University); P30CA060553 (NIH)
Record Dates: First submitted 2024-05-06; First posted 2024-05-13 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Recurrent Glioblastoma, IDH-Wildtype; Recurrent WHO Grade 2 Glioma; Recurrent WHO Grade 3 Glioma; Recurrent WHO Grade 4 Glioma
MeSH Terms: conditions — Glioblastoma | interventions — Specimen Handling; Magnetic Resonance Spectroscopy; Temozolomide; 3-aminopyridine-2-carboxaldehyde thiosemicarbazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 3 (triapine, surgical resection, temozolomide) (Experimental): Patients receive triapine PO QD for 5 days prior to surgical resection. After surgical resection, patients receive temozolomide PO QD and triapine PO QD on days 1-5 of each cycle. Treatment repeats every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo MRI at screening and on study and undergo collection of blood samples on study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Magnetic Resonance Imaging; Other: Questionnaire Administration; Procedure: Resection; Drug: Temozolomide; Drug: Triapine
- Groups 1 and 2 (temozolomide, triapine) (Experimental): Patients receive temozolomide PO QD and triapine PO QD on days 1-5 of each cycle. Treatment repeats every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo MRI at screening and on study and undergo collection of blood samples on study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Magnetic Resonance Imaging; Other: Questionnaire Administration; Drug: Temozolomide; Drug: Triapine

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Other: Questionnaire Administration — Ancillary studies
Procedure: Resection — Undergo surgical resection
  Other Names: Surgical Resection
  Arms: Group 3 (triapine, surgical resection, temozolomide)
Drug: Temozolomide — Given PO
  Other Names: CCRG-81045; Gliotem; Imidazo[5,1-d]-1,2,3,5-tetrazine-8-carboxamide, 3, 4-dihydro-3-methyl-4-oxo-; M & B 39831; M and B 39831; Methazolastone; RP-46161; SCH 52365; Temcad; Temizole; Temodal; Temodar; Temomedac; TMZ
Drug: Triapine — Given PO
  Other Names: 3-aminopyridine-2-carboxaldehyde thiosemicarbazone; 3-AP; 3-Apct; OCX-0191; OCX-191; OCX191; PAN-811

SUMMARY:
This phase I trial tests the safety, side effects, and best dose of triapine in combination with temozolomide in treating patients with glioblastoma that has come back after a period of improvement (recurrent). Triapine inhibits an enzyme responsible for producing molecules required for the production of deoxyribonucleic acid (DNA), which may inhibit tumor cell growth. Temozolomide is in a class of medications called alkylating agents. It works by damaging the cell's DNA and may kill tumor cells and slow down or stop tumor growth. Giving triapine in combination with temozolomide may be safe, tolerable, and/or effective in treating patients with recurrent glioblastoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the recommended phase 2 dose (RP2D) for triapine (3-AP) in combination with temozolomide (TMZ).

SECONDARY OBJECTIVES:

I. To evaluate the safety profile of triapine in combination with temozolomide (TMZ).

II. To evaluate progression-free survival (PFS). III. To evaluate overall survival (OS). IV. To evaluate the overall response rate (ORR) per Response Assessment in Neuro-Oncology (RANO) criteria.

EXPLORATORY OBJECTIVES:

I. To investigate the distribution of triapine within tumor and peritumoral areas post oral administration and correlation with serum levels.

II. To investigate the potential interaction of drug absorption when administrating oral triapine and temozolomide together by measuring plasma levels triapine and temozolomide post administration.

III. To evaluate oral triapine plasma pharmacokinetics and corresponding methemoglobin level by venous blood gas proportion.

IV. To evaluate the quality of life per Functional Assessment of Cancer Therapy-Brain (FACT-Br) for patients treated with triapine and temozolomide.

OUTLINE: This is a dose-escalation study of triapine in combination with temozolomide. Patients with recurrent glioblastoma not planning to undergo surgery are assigned to group 1 or group 2. Patients with recurrent glioblastoma planning to undergo surgery are assigned to group 3.

GROUPS 1 AND 2: Patients receive temozolomide orally (PO) once daily (QD) and triapine PO QD on days 1-5 of each cycle. Treatment repeats every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo magnetic resonance imaging (MRI) at screening and on study and undergo collection of blood samples on study.

GROUP 3: Patients receive triapine PO QD for 5 days prior to surgical resection. After surgical resection, patients receive temozolomide PO QD and triapine PO QD on days 1-5 of each cycle. Treatment repeats every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo MRI at screening and on study and undergo collection of blood samples on study.

After completion of study treatment, patients are followed up at 30 days and then every 3 months for up to 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed World Health Organization (WHO) grade 2-4 glioma, isocitrate dehydrogenase (IDH) wild type (WT) (by immunohistochemistry [IHC] R132H negative [neg] or sequencing). Astrocytoma with molecular features of glioblastoma (GBM). Confirmed diagnosis via molecular testing
* Patients must have an established diagnosis of recurrent glioblastoma and:

  * Group 1 and 2: recurrent glioblastoma
  * Group 3: Surgically amenable recurrent glioblastoma
* Patients must have stable or decreasing dose of corticosteroids equivalent to ≤ 6 mg dexamethasone, for ≥ 7 days prior to registration
* Patients with disease that has progressed after a standard or investigational first-line therapy (e.g. radiotherapy [RT], RT plus temozolomide) with or without tumor treating fields therapy (TTFields)

  * Note: Patients who have received fractionated first-line radiation therapy and no prior chemotherapy (e.g. as common practice for MGMT unmethylated tumors), or who have participated in an investigational protocol substituting TMZ for a novel agent are eligible
* Patients must be able to undergo contrast-enhanced magnetic resonance imaging (MRI)
* Patients must be age ≥ 18 years
* Patients must exhibit a Karnofsky performance status ≥ 70
* Leukocytes (white blood cells [WBC]) ≥ 3,000/mcL
* Absolute neutrophil count (ANC) ≥ 1,500/mcL
* Hemoglobin (Hgb) ≥ 8 g/dL (transfusion may be used for eligibility outside of 7 days)
* Platelets (PLT) ≥ 100,000/mcL (transfusion or growth factor may be used for eligibility outside of 7 days)
* Total bilirubin ≤ 2 x institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) ≤ 3 x institutional ULN
* Creatinine ≤ 1.5 x institutional ULN
* International normalized ratio (INR) ≤ 1.5 x ULN
* Prothrombin time (PT)/partial thromboplastin time (PTT) ≤ 1.5 x ULN
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better
* Patients of child-bearing potential (POCBP) must agree to use two forms of adequate contraception (hormonal or barrier method of birth control, abstinence) from time of informed consent and for the duration of study participation. Patients who can impregnate their partners must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) from time of informed consent and for the duration of study participation

  * Should a patient become pregnant or suspect they are pregnant while they or their partner is participating in this study, they should inform their treating physician immediately.
  * Note: At the discretion of the investigator, acceptable methods of contraception may include total abstinence in cases where the lifestyle of the patient ensures compliance. (Periodic abstinence [e.g., calendar, ovulation, symptothermal, postovulation methods] and withdrawal are not acceptable methods of contraception.)
  * Note: A POCBP is any person with an egg-producing reproductive tract (regardless of gender, sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

    * Has not undergone a hysterectomy, bilateral salpingectomy, or bilateral oophorectomy
    * Has had menses at any time in the preceding 12 consecutive months (and therefore has not been naturally postmenopausal for > 12 months) (in patients > 45 years of age in the absence of other biological or physiological causes)

      * Potential POCBP who may be menopausal and are < 55 years of age must have a serum follicle-stimulating hormone (FSH) level > 40 mIU/mL to confirm menopause
      * Note: Documentation may include review of medical records, medical examination, or medical history interview by study site staff
* Patient must be willing and able to comply with the protocol for the duration of the study and provide written, signed, and dated informed consent prior to study registration.

  * NOTE: No study-specific screening procedures may be performed until written consent has been obtained
* Patients must have the ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have a prior or concurrent malignancy that may interfere with study treatment or safety

  * NOTE: Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible, per principal investigator (PI) discretion
* Patients who are receiving any other investigational agents.

  * Exceptions: COVID-19 vaccine and treatment is allowed, per PI's discretion
* Patient's interval since last cytotoxic therapy ≥ 1 cycle or ≥ 2 biological half-lives, i.e.

  * ≥ 28 days since start of last cycle of temozolomide (cycle length-28 days)
  * ≥ 42 days since start of last cycle of lomustine or other nitrosourea (cycle length-42 days)
  * ≥ 21 days since start of last cycle of a small molecule targeted agent (cycle length-21 days)
  * ≥ 42 days from last bevacizumab infusion (cycle length-42 days)
* Patients who have a history of allergic reactions attributed to compounds of similar chemical composition to temozolomide or triapine
* Patients with spinal cord and diffuse leptomeningeal dissemination
* Patients with a history of G6PD deficiency or other congenital or autoimmune hemolytic disorders. All participants will be screened for G6PD levels prior to registration
* Patients who have an uncontrolled intercurrent illness including, but not limited to any of the following:

  * Have uncontrolled epilepsy
  * Have an uncontrolled intercurrent illness
  * Are pregnant or nursing
  * Concurrent malignancy (outside of glioblastoma) that requires tumor directed treatment
  * Known concurrent shingles, herpes, cytomegalovirus (CMV) infection
  * Known concurrent opportunistic fungal infection
  * Known immunodeficiency that could lead to opportunistic infections
  * Psychiatric illness/social situations that would limit compliance with study requirements
  * Any other illness or condition that the treating investigator feels would interfere with study compliance or would compromise the patient's safety or study endpoints
* Patients who are pregnant or nursing. Pregnant patients are excluded from this study because temozolomide is an alkylating agent with potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with temozolomide, breastfeeding should be discontinued if the mother is treated with temozolomide
* Patients who are unable to swallow oral medication or have problems/diseases that affect absorption or oral medication
* Patients with a known history of human immunodeficiency virus (HIV), hepatitis B virus (HBV), and/or hepatitis C virus (HCV). If patient does not have a known history testing will not be conducted

  * Note: Temozolomide is an immunosuppressive agent. Patients with a known history of HIV, HBV, and HCV, and unexplained opportunistic infections are not eligible due to safety reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-07-23 (Actual); Primary Completion 2029-05-12 (Estimated); Study Completion 2030-05-12 (Estimated)

PRIMARY OUTCOMES:
Recommended phase 2 dose for triapine in combination with temozolomide | At the end of Cycle 1 (each cycle is 28 days) + 7 days (up to cycle 2 day 7)
  The recommended phase 2 dose will be based on treatment-emergent and drug-related toxicity. Dose limiting toxicities and adverse events (AEs) will be assessed by Common Terminology Criteria for Adverse Events (CTCAE) version (v.) 5.0.

SECONDARY OUTCOMES:
Incidence of AEs and serious AEs | Up to 30 days after last administration of study drug
  Will evaluate the occurrence of toxicity (AEs and serious AEs) and the number of patients who discontinue treatment due to toxicity. Toxicity will be assessed by CTCAE v. 5.0. Adverse events will be sorted (by type, severity [grade], timing, and attribution to triapine), collected, and reported according to CTCAE v5.0.
Progression free survival (PFS) | From baseline until the patient experiences disease progression, initiates subsequent anti-cancer therapy, completes study participation, or experiences death from any cause, assessed at 6, 12, and 24 months
  Progression will be determined by clinical progression or by radiographic imaging as assessed by Response Assessment in Neuro-Oncology (RANO) criteria. The median and corresponding 95% confidence interval will also be estimated.
Overall survival | From time of diagnosis until the patient initiates subsequent anti-cancer therapy, completes study participation, or experiences death from any cause, assessed at 6, 12, and 24 months
  Will be described by Kaplan-Meier curve. The median and corresponding 95% confidence interval will also be estimated.
Overall response rate (ORR) | From baseline until the response has been confirmed, the patient experiences disease progression, the patient initiates, subsequent anti-cancer therapy, or the patient completes study participation, assessed up to 24 months
  ORR will be assessed by RANO criteria. To determine the ORR, this endpoint will calculate the proportion of treated patients who experience an overall response (complete response [CR] or partial response [PR] per RANO criteria). The date of first response for either CR or PR will be used for the calculation of ORR. Will be estimated using the expansion cohort, along with its 95% confidence interval.

CONTACTS AND LOCATIONS:
Overall Officials: Karan Dixit, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States